CLINICAL TRIAL: NCT00190918
Title: A Phase II Trial of Pemetrexed (Alimta) in the Treatment of Recurrent or Persistent Low Risk Gestational Trophoblastic Tumor
Brief Title: A Trial for Patients With Gestational Trophoblastic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Gynecologic Oncology Group (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8366; H3E-US-JMGR
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-08

CONDITIONS: Trophoblastic Neoplasms; Uterine Neoplasms; Hydatidiform Mole; Choriocarcinoma
MeSH Terms: conditions — Trophoblastic Neoplasms; Uterine Neoplasms; Hydatidiform Mole; Choriocarcinoma | interventions — Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed

SUMMARY:
This phase II study is evaluating the activity of Pemetrexed in patients diagnosed with low risk Gestational Trophoblastic Tumor (GTT) that have failed prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or recurrent low risk Gestational Trophoblastic Tumor (GTT)
* WHO score 2-6 (re-evaluated at the time of relapse
* Histologically confirmed complete or partial moles on initial evacuation
* Patients with mild to moderate renal insufficiency should avoid taking NSAIDs with short elimination half-lives for a period of 2 days before, the day of, and 2 days following administration of pemetrexed.
* All patients taking NSAIDs with longer half-lives, should interrupt dosing for at least 5 days before, the day of, and 2 days following pemetrexed administration.
* Folic Acid (350-1000 micrograms) must be given daily beginning approximately 5-7 days prior to first dose of pemetrexed and continuing daily until 3 weeks after the last dose of study therapy.
* Vitamin B12 (1000 micrograms) will be administered as an intramuscular injection approximately 1 to 2 weeks prior to first dose of pemetrexed and repeated approximately every 9 weeks until 3 weeks after the last dose of study therapy.

Exclusion Criteria:

* Previous treatment that included chemotherapy other than actinomycin -D or methotrexate (+/- folinic acid).
* Patients with more than 8 metastatic lesions identified
* Patients with metastases to liver, spleen, brain, kidney or GI tract

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To determine the activity of Pemetrexed in failed low risk Gestational Trophoblastic Tumor (GTT) patients

SECONDARY OUTCOMES:
To determine the toxicity of Pemetrexed in failed low risk Gestational Trophoblastic Tumor (GTT) patients

CONTACTS AND LOCATIONS:
Overall Officials: David Miller, MD, Study Chair — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group 215-854-0770, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com